CLINICAL TRIAL: NCT07102381
Title: A Phase 2, Randomized, Multicenter, Open-label Neoadjuvant Study Evaluating Zanidatamab in Combination With Chemotherapy in Participants With HER2-positive Breast Cancer
Brief Title: A Phase 2 Neoadjuvant Study of Zanidatamab in Combination With Chemotherapy in Participants With HER2-positive Breast Cancer
Acronym: EmpowHER 208
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Jazz Pharmaceuticals Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JZP598-208; 2025-523204-68-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: HER2-positive Breast Cancer; Breast Cancer
Keywords: HER2-positive early breast cancer; invasive breast carcinoma; zanidatamab; breast neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — zanidatamab; Paclitaxel; Docetaxel; Carboplatin; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Zanidatamab with paclitaxel (Active Comparator): Zanidatamab in combination with chemotherapy paclitaxel
  Interventions: Drug: Zanidatamab; Drug: Paclitaxel
- Zanidatamab with docetaxel and carboplatin (Active Comparator): Zanidatamab in combination with chemotherapy docetaxel and carboplatin
  Interventions: Drug: Zanidatamab; Drug: Docetaxel; Drug: Carboplatin
- Trastuzumab and pertuzumab with docetaxel and carboplatin (Active Comparator): Trastuzumab and pertuzumab in combination with chemotherapy docetaxel and carboplatin
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Zanidatamab — Administered intravenously (IV)
  Other Names: ZW25; JZP598; ZIIHERA®
  Arms: Zanidatamab with docetaxel and carboplatin; Zanidatamab with paclitaxel
Drug: Paclitaxel — Administered intravenously (IV)
  Arms: Zanidatamab with paclitaxel
Drug: Docetaxel — Administered intravenously (IV)
  Arms: Trastuzumab and pertuzumab with docetaxel and carboplatin; Zanidatamab with docetaxel and carboplatin
Drug: Carboplatin — Administered intravenously (IV)
  Arms: Trastuzumab and pertuzumab with docetaxel and carboplatin; Zanidatamab with docetaxel and carboplatin
Drug: Trastuzumab — Administered intravenously (IV)
  Arms: Trastuzumab and pertuzumab with docetaxel and carboplatin
Drug: Pertuzumab — Administered intravenously (IV)
  Arms: Trastuzumab and pertuzumab with docetaxel and carboplatin

SUMMARY:
The purpose of this study is to see if zanidatamab is safe and effective, when combined with chemotherapy, in treating people who has Human Epidermal Growth Factor Receptor 2 (HER2)-positive, early-stage breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Has Stage II or III histologically confirmed invasive breast carcinoma.
2. Has histologically confirmed HER2-positive breast cancer
3. Has a known hormone receptor (HR) status of the primary tumor
4. Participants with multifocal or multicentric disease are eligible if the largest tumor (which must be larger than or equal to 2 cm in diameter) is HER2-positive, and the treating physician has determined the participant should be treated as HER2-positive.
5. Agrees to undergo a mastectomy or breast conserving surgery (BCS) after neoadjuvant therapy.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate organ function
8. Has an LVEF ≥ 50% as determined by either ECHO or MUGA obtained within 4 weeks prior to first dose of study intervention.
9. Adequate contraceptive precautions

Exclusion Criteria:

1. Has Stage IV (metastatic) breast cancer.
2. Has bilateral breast cancer.
3. Has a history of any severe and/or uncontrolled medical conditions or other conditions that, in the opinion of the investigator, could affect the participant's involvement in the study.
4. Has uncontrolled hypertension
5. Has significant symptoms from peripheral neuropathy
6. Has an active uncontrolled infection
7. Has a history of life-threatening hypersensitivity to monoclonal antibodies or to recombinant proteins or excipients in the drug formulation of zanidatamab or other study interventions.
8. Known active hepatitis B or C infection.
9. Has another malignancy diagnosed within the last 5 years. Exceptions include previously treated non melanomatous skin cancers, carcinoma in-situ, and melanoma in-situ.
10. Was treated with chemotherapy, anti-HER2 therapy, radiation therapy, endocrine therapy, or experimental therapy for invasive breast cancer
11. Is planning to receive concurrent therapy with any other investigational agent or anti-cancer therapy not specified in the protocol
12. Receipt of a live vaccine within 4 weeks prior to enrollment
13. Has a known hypersensitivity to any components of the study interventions, including chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with pCR | Up to 8 months
  Pathologic complete response (pCR) is defined as lacking all signs of cancer in the tissue samples removed in the breast or axilla (armpit) during surgery or biopsy after study treatment

SECONDARY OUTCOMES:
Number of participants with Pathologic response by Residual Cancer Burden (RCB) classification | Up to 8 months
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 23 months
Number of Participants Discontinuing Study Treatment Due to TEAEs | Up to 23 months
Number of participants that completed breast conservation surgery (BCS) | Up to 8 months
Event Free Survival (EFS) | Up to 46 months
  EFS is defined as the time (in months) from randomization to disease progression, disease recurrence, or death from any cause
Overall Survival (OS) | Up to 46 months
  OS is defined as the time in months from randomization to the date of death due to any cause.
Number of participants reporting Symptomatic Adverse Events based on Patient-reported Outcome-Common Terminology Criteria for AEs (PRO-CTCAE) | Up to 23 months
  Symptomatic AEs assessed by the PRO-CTCAE are analyzed at the item level with symptom severity, frequency, and interference scored from 0 to 4 and presence/absence scored 0 to 1, and higher scores reflect worse symptoms.
Number of participants reporting Symptomatic Adverse Events based on European Organisation for Research and Treatment of Cancer (EORTC) Item Library | Up to 23 months
  Symptomatic AEs assessed by the EORTC Item Library Forms are analyzed at the item level with scores ranging from 1 to 4, where a 4 indicates more severe symptoms.
Percentage of all treated participants reporting overall side-effect bother on the Functional Assessment of Chronic Illness Therapy General Physical Item 5 (FACIT-GP5) | Up to 23 months
  The Functional Assessment of Chronic Illness Therapy (FACIT) GP5 Item score ranges from 0 (Not at all) to 4 (Very Much), where higher scores reflect greater bother from treatment side effects.
Serum Concentrations of Zanidatamab | Up to 18 months
Number of Participants Positive for Anti-drug Antibodies to Zanidatamab | Up to 18 months

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - The Oncology Institute, Lakeland, Florida
  - Accellacare of McFarland, Ames, Iowa
  - LSU Health Sciences Center, Shreveport, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - Maryland Oncology Hematology, Laurel, Maryland
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Astera Cancer Care (Formerly Regional Cancer Care Associates), East Brunswick, New Jersey
  - Medical Oncology Hematology Associates, Newark, New Jersey
  - Hematology Oncology Associates of Central New York, Camillus, New York
  - Sarah Cannon Research Institute (Nashville), Nashville, Tennessee
  - Texas Oncology DFW, Dallas, Texas
  - Texas Oncology Gulf Coast, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Shenandoah Oncology, Winchester, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com.
URL: https://www.jazzpharma.com/science/clinical-trial-data-sharing